CLINICAL TRIAL: NCT06696820
Title: Efficacy and Safety of Early Combined Therapy with PCSK9 Inhibitors and Statins in Acute Ischemic Stroke (CAPTAIN)--A Multicenter, Prospective, Randomized Trial
Brief Title: Efficacy and Safety of Early Combined Therapy with PCSK9 Inhibitors and Statins in Acute Ischemic Stroke
Acronym: CAPTAIN
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Xiang Luo (Other)
Collaborators: The Third People's Hospital of Hubei Province (Other); Hubei Shiyan People's Hospital (Unknown); Yichang Central People's Hospital (Other); The Fifth Hospital of Wuhan (Other); Shanghai Zhongshan Hospital (Other); Renmin Hospital of Wuhan University (Other); Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other); Wuhan Third Hospital (Other); Taihe Hospital (Other); Suizhou Hospital, Hubei University of Medicine (Unknown); Hubei Xinhua Hospital (Other); Tianyou Hospital Affiliated to Wuhan University of Science and Technology (Other); Minda Hospital Affiliated to Hubei University for Nationalities (Unknown)
Responsible Party: Sponsor-Investigator, Xiang Luo, Principal Investigator, Tongji Hospital
Organization: Tongji Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 1100939
Record Dates: First submitted 2024-11-17; First posted 2024-11-20 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2024-11

CONDITIONS: Acute Ischemic Stroke
Keywords: Acute Ischemic Stroke; PCSK9 inhibitor
MeSH Terms: conditions — Ischemic Stroke | interventions — Atorvastatin; Rosuvastatin Calcium

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- PCSK9 inhibitors combined with atorvastatin/rosuvastatin (Experimental)
  Interventions: Drug: PCSK9 inhibitors combined with atorvastatin/rosuvastatin
- Atorvastatin/rosuvastatin (Sham Comparator)
  Interventions: Drug: Atorvastatin/Rosuvastatin

INTERVENTIONS:
Drug: PCSK9 inhibitors combined with atorvastatin/rosuvastatin — A single subcutaneous injection of 420 mg Iroceliumab upon admission, along with a standard dose of 20 mg Atorvastatin or 10 mg Rosuvastatin
  Other Names: 222
  Arms: PCSK9 inhibitors combined with atorvastatin/rosuvastatin
Drug: Atorvastatin/Rosuvastatin — Conventional Atorvastatin 20 mg / Rosuvastatin 10 mg
  Arms: Atorvastatin/rosuvastatin

SUMMARY:
This study is an investigator-initiated, multicenter, prospective, open-label, endpoint-blinded, randomized controlled trial (PROBE design) that includes patients with moderate or severe symptomatic intracranial large vessel atherosclerotic stenosis (sICAS) who present with acute ischemic stroke within 48 hours of symptom onset.

Patients will be centrally randomized in a 1:1 ratio into two groups:

Experimental Group: A single subcutaneous injection of 420 mg evolocumab upon admission, combined with standard doses of atorvastatin 20 mg or rosuvastatin 10 mg, along with other standard guideline-based medical treatments.

Control Group: Standard doses of atorvastatin 20 mg or rosuvastatin 10 mg, with the remainder of treatment based on current guidelines.

The primary objective of the study is to evaluate whether early combination therapy with a PCSK9 inhibitor and statins within 48 hours of symptom onset can reduce the incidence of early neurological deterioration in patients with symptomatic intracranial atherosclerotic stenosis (sICAS). The secondary objectives include comparing the effects of early PCSK9 inhibitor and statin combination therapy versus statin monotherapy on the 90-day neurological outcomes of AIS patients, improving early neurological recovery, and reducing the recurrence rate of stroke at 30 and 90 days. The safety objective is to assess whether the combination of early PCSK9 inhibitors and statins, compared to statin monotherapy, increases the incidence of moderate-to-severe systemic bleeding within 3 days post-randomization (based on the GUSTO scale), any type of intracranial hemorrhage (according to the ECASS III criteria), and all-cause mortality within 90 days.

DETAILED DESCRIPTION:
Acute ischemic stroke (AIS) is a cerebrovascular disease with high incidence, recurrence, and disability rates, posing a serious threat to human health. Symptomatic intracranial atherosclerotic stenosis (ICAS) is one of the most common causes of ischemic stroke globally. In Asian populations, ICAS is the predominant subtype, accounting for approximately 50% of all ischemic strokes. Despite aggressive and standardized medical therapy, patients with ICAS still face a high recurrence rate of stroke and incidence of early neurological deterioration (END). Over 50% of cases of END occur within 72 hours of AIS onset and are defined as an increase in the NIHSS score by ≥2 or 4 points from baseline, which is closely linked to clinical outcomes. Two previous randomized controlled trials (RCTs) found that combined clopidogrel and aspirin dual antiplatelet therapy can prevent END and improve neurological outcomes in AIS patients. However, the occurrence of END remains high, as drug resistance and swallowing difficulties may hinder timely administration.

Multiple RCTs have shown that statin therapy can reduce the risk of recurrent stroke and improve neurological outcomes, and it is consistently recommended by both domestic and international ischemic stroke guidelines. The SPARCL study, published in the New England Journal of Medicine, demonstrated that in patients with a history of recent stroke, lowering LDL-C from ≥2.6 mmol/L to <1.8 mmol/L significantly reduces the risk of recurrent stroke and cardiovascular events. More recently, the INSPIRES study, published in JAMA Neurology, indicated that early statin therapy within 3 days of AIS onset significantly reduces adverse neurological outcomes, such as the proportion of patients with a 90-day mRS score of 2-6 (11.4% vs. 9.8%, P<0.05), compared to delayed statin therapy, although no significant difference was observed in recurrent stroke events within 90 days. As stroke guidelines have evolved, the LDL-C target for secondary prevention has been lowered from 2.6 mmol/L to below 1.8 mmol/L. Statins and other lipid-lowering agents work through different mechanisms affecting cholesterol synthesis, absorption, and clearance, and their combined use can produce a synergistic effect. At the 2024 annual meeting of the Chinese Stroke Society, experts proposed a new concept for lipid management in AIS patients, focusing on residual lipid risk and early combination therapy to achieve more rapid, sustained, and stable lipid control.

Proprotein convertase subtilisin/kexin type 9 (PCSK9) inhibitors are a novel class of monoclonal antibody-based lipid-lowering drugs that reduce serum LDL-C levels by inhibiting the binding of PCSK9 to LDL receptors. PCSK9 inhibitors are highly effective in lowering lipid levels with minimal adverse effects and high safety. The main PCSK9 inhibitors approved for clinical use are alirocumab and evolocumab. Recent international guidelines have clearly stated that PCSK9 inhibitors can be used in combination with statins or other lipid-lowering agents or as monotherapy in patients who are statin-intolerant or for whom statins are contraindicated. Due to the complementary mechanisms of action between statins and PCSK9 inhibitors, their combined use has been shown to provide a greater-than-additive lipid-lowering effect. Post-hoc analyses of the FOURIER study, published in Stroke, and the ODYSSEY study, published in Circulation, confirmed that in patients with atherosclerotic cardiovascular disease, combination therapy with statins and PCSK9 inhibitors significantly reduced the risk of ischemic stroke (1.2% vs. 1.5%, P=0.005; 1.2% vs. 1.6%, P=0.01), with no significant difference in the risk of hemorrhagic stroke between the groups.

However, it remains unclear whether the combination of statins and PCSK9 inhibitors improves neurological outcomes in acute ischemic stroke, particularly in patients with ICAS, as high-quality evidence is lacking. A multicenter, prospective cohort study found that for AIS patients with ICAS, early combination therapy with statins and PCSK9 inhibitors within 7 days of onset significantly reduced the risk of early stroke recurrence within 30 days (5.59% vs. 2.16%, P=0.039). A single-center, retrospective cohort study demonstrated that early combination therapy with statins and PCSK9 inhibitors within 24 hours of stroke onset significantly reduced the incidence of early neurological deterioration (increase in NIHSS score ≥2 points) within 72 hours compared to statin monotherapy (31.9% vs. 12.5%, P=0.005). Another single-center, retrospective cohort study found that for AIS patients undergoing thrombectomy, early combination therapy with statins and PCSK9 inhibitors reduced the proportion of patients with an NIHSS score at discharge and an mRS score of ≤3 (35.6% vs. 52.4%, P=0.041) without increasing the risk of symptomatic intracranial hemorrhage (8.7% vs. 2.4%, P=0.16). Although the reduction in early neurological deterioration was not statistically significant (20.1% vs. 11.9%, P=0.21), these studies support the effectiveness and safety of statin and PCSK9 inhibitor combination therapy in improving neurological outcomes in AIS, providing a reliable foundation for further high-quality RCTs.

This multicenter, prospective, randomized controlled study aims to investigate and evaluate the effects of early combination therapy with PCSK9 inhibitors and statins on early neurological deterioration and other neurological outcome measures in patients with symptomatic intracranial atherosclerotic stenosis, which holds significant clinical value.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Acute ischemic stroke diagnosed by CT or MRI of the head.
3. Symptom onset to randomization within 48 hours, including wake-up strokes or strokes without a witnessed onset. The time of symptom onset is defined as the "last known normal time."
4. NIHSS score ≤ 20.
5. mRS score of 0-1 prior to the current stroke.
6. Moderate or severe intracranial stenosis or occlusion (≥50%) confirmed by CTA, MRA, or DSA, involving the responsible intracranial arteries: intradural internal carotid artery, M1-2 segments of the middle cerebral artery, A1 segment of the anterior cerebral artery, V4 segment of the vertebral artery, basilar artery, or P1 segment of the posterior cerebral artery.
7. The participant or legal representative has signed the informed consent form.

Exclusion Criteria:

1. Cardiogenic embolism (e.g., atrial fibrillation, cardiac valvular disease, etc.).
2. Symptomatic intracranial stenosis or occlusion due to arteritis, arterial dissection, moyamoya disease, or other similar conditions.
3. Patients who have received intravenous thrombolysis or mechanical thrombectomy.
4. Use of PCSK9 inhibitors within the 1 month prior to the onset of the stroke.
5. Allergy to statins or PCSK9 inhibitors.
6. Active liver disease, including unexplained persistent elevations of alanine aminotransferase (ALT) and/or aspartate aminotransferase (AST).
7. Known severe renal impairment (creatinine clearance <30 mL/min).
8. Myopathy.
9. Concurrent use of cyclosporine.
10. Known pregnancy or breastfeeding, or a positive pregnancy test prior to randomization.
11. Life expectancy <3 months (e.g., due to severe cardiopulmonary disease, renal failure, malignancy, or other terminal conditions).
12. Participation in other interventional clinical trials that may impact outcome assessments.
13. Any other condition that, in the investigator's judgment, makes the patient unsuitable for participation or poses significant risks to the patient.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 416 (Estimated)
Dates: Start 2024-11-29 (Actual); Primary Completion 2027-06-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Proportion of early neurological deterioration | Within 3 days of randomization
  The proportion of patients with an increase of ≥2 points in the NIHSS score from baseline within 3 days post-randomization
The proportion of moderate-to-severe systemic bleeding within 3 days post-randomization (according to the GUSTO criteria) | Within 3 days of randomization

SECONDARY OUTCOMES:
ProportioThe proportion of patients with an increase of ≥4 points in the NIHSS score from baseline within 3 days post-randomizationn of early neurological improvement | Within 3 days of randomization
Proportion of early neurological improvement | Within 3 days of randomization
  The proportion of patients with a reduction of ≥4 points in the NIHSS score from baseline or a score reduced to 0-1 within 3 days post-randomization.
The change in NIHSS score from baseline to 1 day post-randomization. | One day after randomization
The change in NIHSS score from baseline to 3 day post-randomization. | 3 day after randomization
The change in NIHSS score from baseline to 7 day post-randomization. | 7 days after randomization
mRS score at 90 days post-randomization | 90 days after randomization
Stroke recurrence rate within 30 days post-randomization | Within 30 days of randomization
Stroke recurrence rate within 90 days post-randomization | Within 90 days of randomization
The change in lipid parameters from baseline to 7 days post-randomization or at discharge | 7 days after randomization
The proportion of systemic bleeding within 3 days post-randomization (according to the GUSTO criteria) | Within 3 days of randomization
The proportion of any type of intracranial hemorrhage within 3 days post-randomization (according to the ECASS III criteria) | Within 3 days of randomization
The incidence of any adverse events or serious adverse events within 90 days post-randomization | Within 90 days of randomization
All-cause mortality rate within 90 days post-randomization | Within 90 days of randomization

CONTACTS AND LOCATIONS:
Locations (2):
- China (2):
  - Tongji Hospital, Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei
  - Tongji Hospital,Tongji Medical College, Huazhong University of Science and Technology, Wuhan, Hubei

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gutierrez J, Turan TN, Hoh BL, Chimowitz MI. Intracranial atherosclerotic stenosis: risk factors, diagnosis, and treatment. Lancet Neurol. 2022 Apr;21(4):355-368. doi: 10.1016/S1474-4422(21)00376-8. Epub 2022 Feb 7. PMID 35143758